CLINICAL TRIAL: NCT03382041
Title: Intramedullary Nailing of Tibia Shaft Fractures With Carbon Fiber Implants Versus Titanium Nails: A Randomized Cohort Study
Brief Title: Carbon Fiber Implants
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Original PI no longer works at UAB
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: CarboFix Orthopedics (Industry)
Responsible Party: Principal Investigator, Clay Spitler, Primary Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: F160824002
Record Dates: First submitted 2017-11-13; First posted 2017-12-22 (Actual); Results first posted 2022-03-02 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Tibial Shaft Fractures

STUDY DESIGN:
Intervention Model Description: The investigators will compare intramedullary nailing( placing a rod in the tibia) of open and closed tibia shaft fractures with carbon fiber implant (tibial nail) versus titanium implant (tibial nail) in a Level I trauma setting.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Carbon Fiber Implant (Experimental): There is an alternative to the standard treatment, which is carbon fiber implants (tibial nails), especially in the prophylactic reinforcement of bones susceptible to pathological fractures following metastatic tumors. The new carbon fiber has also been used in the treatment of tibial non-union (non- healing bone); which has shown satisfactory outcomes.
  Interventions: Device: Carbon Fiber Implant
- Titanium Implant (Active Comparator): The standard of practice in the treatment of fractures of the tibial shaft and other long bones has been the intramedullary nailing using titanium or stainless steel implants.
  Interventions: Device: Titanium Implant

INTERVENTIONS:
Device: Carbon Fiber Implant — A cannulated rod, made of long carbon fiber reinforced polymer, with interlocking holes at its proximal and distal ends. The Nail provides for a slight bend. A Tantalum radiopaque marker along the Nail longitudinal axis provides for its visualization under fluoroscopy. The Nail proximal end is marked by a tantalum marker.
  Arms: Carbon Fiber Implant
Device: Titanium Implant — An intramedullary rod, also known as an intramedullary nail (IM nail) or inter-locking nail or Küntscher nail (without proximal or distal fixation), is a metal rod forced into the medullary cavity of a bone. IM nails have long been used to treat fractures of long bones of the body
  Arms: Titanium Implant

SUMMARY:
The investigators will compare intramedullary nailing of open and closed tibia shaft fractures with carbon fiber implant versus titanium implant in a Level I trauma setting.

DETAILED DESCRIPTION:
The tibia (long bone in the leg) bears most of the body weight and is the most commonly fractured long bone in the body. According to the National Center for Health Statistics; tibia, fibula and ankle fractures account for an annual sum of 581,000 fractures. Of all long bone fractures, the tibia is the most common site for non -union(failure to heal).

For many years, the standard practice in the treatment of fractures of the tibia shaft and other long bones has been intramedullary nailing (placing rod in the bone)using titanium or stainless steel implants( tibial nails).

More recently however, orthopaedic surgeons have found an alternative to the standard carbon fiber implants (tibial nails), especially in the prophylactic reinforcement of bones susceptible to pathological fractures following metastatic tumors. The new carbon fiber has also been used in the treatment of tibial non-union (non- healing bone); which has shown satisfactory outcomes. A clear advantage over titanium implants (tibial nails) is the carbon fiber's radiolucent (ability to see through the implant on x-ray) property. This allows for improved visualization of early healing and the reduction of fracture segments (i.e. fracture alignment) without the typical radiopaque (inability to see through the implant on x-ray) density and artifact found with metals on x-ray, MRI or CT Scans. The early visualization of callus formation8(healing) may therefore serve as a good prognostic predictor of successful union.

Thus orthopaedic trauma patients, especially in cases of polytrauma may heal faster; attain earlier weight bearing status, and independence, decrease rehabilitation center stays and advance recovery with possible quicker return to work. These benefits have economic significance in reducing direct costs to patients and their families as well as to the healthcare system. Use of carbon fiber implants (tibial nails) seems to hold the promise of a shorter recovery time with better functional outcome than with more rigid titanium implants (tibial nails). This is due to the carbon fiber implants(tibial nails) elasticity (flexibility) which is close to that of bone, preventing excessive rigidity and possible non- union (non -healing bone).

Intramedullary nails have continued to evolve, beginning with stainless steel implants and progressing to titanium. The titanium nail has been used over several years and the carbon fiber is a newer material and is now used by several institutions for treatment of tibial shaft fractures. There are no studies that directly compare the two nails in a prospective manner.

The standard of care for treatment of tibial shaft fractures is the use of an intramedullary (rod inside the bone) implant. Both implants perform the same function but are made of different materials. Current treatment of tibia fractures at The University of Alabama at Birmingham (UAB) utilizes both titanium and carbon fiber implants.

ELIGIBILITY:
Inclusion Criteria:

* i. Skeletal maturity (patients included will be 18 - 64 years, i.e. whose epiphyseal/growth plates are closed) ii. Arbeitsgemeinschaft ur Osteosynthesefragen/Orthpaedica Trauma Association (AO/OTA) Fracture class 42; open and closed tibia shaft fracture (Gustilo-Anderson Types I II, and III; Tscherne closed types 0, I, 2 and 3), Tscherne open types I and II.

iii. Fractures amenable to intramedullary nailing (placing a rod within the bone) iv. Fracture gaps less than 2 cm due to bone loss v. In cases of bilateral tibial fractures the investigators would include both if they meet inclusion criteria..

vi. Patient's informed consent or that of a legally acceptable representative

Exclusion Criteria:

i. Subjects currently enrolled in one or more clinical studies ii. Skeletal immaturity (i.e. 17 years and younger) iii. Fractures planned for non-operative management iv. Complex intra-articular involvement of tibia plateau or distal tibia v. Pathologic fractures (fractures secondary to disease) vi. Concomitant ipsilateral tibia shaft fractures with complex pilon and/or plateau fractures requiring fixation vii. Patients already treated or in re-treatment viii. Tibia already infected as diagnosed by the attending physician ix. Patients likely to be lost before completing adequate follow-up, such as prisoners or planned out-of-state (and other likely problems in the investigator's judgment, with maintaining follow-up visit schedule) x. Patient is intellectually challenged or has a severe psychiatric condition xi. Patient is incompetent in the English Language xii. Patient is non-ambulatory before injury or as a consequence of polytrauma xiii. Inability to obtain patient's informed consent and/or that of a legally acceptable representative

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-05-23 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2021-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clay A Spitler, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- The University of Alabama at Birmingham (UAB), Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Carbon Fiber Implant | Titanium Implant
Started | 7 | 13
Completed | 3 | 4
Not Completed | 4 | 9
Not completed — Consent Form Lost | 2 | 1
Not completed — Withdrawal by Subject | 1 | 4
Not completed — Lost to Follow-up | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Carbon Fiber Implant | Titanium Implant | Total
Number analyzed (Participants) | 7 | 13 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 13 | 20
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 5 | 10 | 15
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic | 1 | 0 | 1
  Black | 2 | 4 | 6
  White | 4 | 9 | 13
Region of Enrollment [Number; unit: participants]
  United States | 7 | 13 | 20

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants Identified With Fracture Healing
Description: Will assess radiographically the fracture healing for patients treated with Carbon Fiber and Titanium Implants.
Time Frame: From baseline through 6 weeks.
Population: 7 subjects were withdrawn due to the discretion of the PI, 2 subjects withdrew consent, 6 subjects were lost to follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Carbon Fiber Implant | Titanium Implant
Number analyzed (Participants) | 3 | 4
Participants | 1 | 1

2. Primary Outcome: The Number of Participants Identified With Fracture Healing
Description: Will assess radiographically the fracture healing for patients treated with Carbon Fiber and Titanium Implants.
Time Frame: From baseline through 3 months.
Population: 7 subjects were withdrawn due to the discretion of the PI, 2 subjects withdrew consent, 6 subjects were lost to follow-up, 1 subject did not have x-rays done.
Measure: Count of Participants; unit: Participants
Arm/Group | Carbon Fiber Implant | Titanium Implant
Number analyzed (Participants) | 3 | 3
Participants | 1 | 2

3. Secondary Outcome: Short Musculoskeletal Function Assessment Questionnaire (SMFA).
Description: The SMFA will be administered to patients at 6 months following injury. The scores of dysfunction are calculated by summing up the responses to the items and then transforming the scores according to the formula. This transformation formula gives the final scores which ranged from 0-100. The higher scores indicate poorer function.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Carbon Fiber Implant | Titanium Implant
Number analyzed (Participants) | 3 | 4
units on a scale | 31.53 (20.55) | 38.56 (32.46)

4. Secondary Outcome: Short Musculoskeletal Function Assessment Questionnaire (SMFA) Score.
Description: Patient reported levels of function and satisfaction with the fixation method and overall treatment. The SMFA will be administered to patients at 6 months following injury. The scores of bother are calculated by summing up the responses to the items and then transforming the scores according to the formula. This transformation formula gives the final scores which ranged from 0-100. The higher scores indicate poorer function.
Time Frame: 6 months
Population: One patient wasn't available to evaluate from the Titanium group.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Carbon Fiber Implant | Titanium Implant
Number analyzed (Participants) | 3 | 3
units on a scale | 32.39 (22.60) | 49.24 (46.71)

5. Secondary Outcome: Short Musculoskeletal Function Assessment Questionnaire (SMFA).
Description: Patient reported levels of function and satisfaction with the fixation method and overall treatment. The Short Form Musculoskeletal Assessment (SMFA) will be administered to patients at 12 months following injury. The scores of dysfunction are calculated by summing up the responses to the items and then transforming the scores according to the formula. This transformation formula gives the final scores which ranged from 0-100. The higher scores indicate poorer function.
Time Frame: 12 months.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Carbon Fiber Implant | Titanium Implant
Number analyzed (Participants) | 3 | 4
units on a scale | 29.85 (28.35) | 31.09 (27.85)

6. Secondary Outcome: Short Musculoskeletal Function Assessment Questionnaire (SMFA) Score.
Description: Patient reported levels of function and satisfaction with the fixation method and overall treatment. The Short Form Musculoskeletal Assessment (SMFA) will be administered to patients at 12 months following injury. The scores of bother are calculated by summing up the responses to the items and then transforming the scores according to the formula. This transformation formula gives the final scores which ranged from 0-100. The higher scores indicate poorer function.
Time Frame: 12 months.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Carbon Fiber Implant | Titanium Implant
Number analyzed (Participants) | 3 | 4
units on a scale | 34.09 (32.06) | 37.88 (36.46)

7. Secondary Outcome: Short Musculoskeletal Function Assessment Questionnaire (SMFA) Score.
Description: Patient reported levels of function and satisfaction with the fixation method and overall treatment. The Short Form Musculoskeletal Assessment (SMFA) will be administered to patients at 18 months following injury. The scores of the dysfunction and bother indices are calculated by summing up the responses to the items and then transforming the scores according to the formula. This transformation formula gives the final scores which ranged from 0-100. The higher scores indicate poorer function.
Time Frame: 18 months.
Population: Data was not collected.
Arm/Group | Carbon Fiber Implant | Titanium Implant
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Veterans Rand Health Survey (VR-12)
Description: The Veterans Rand 12 Item Health Survey is a multipurpose, self-administered generic measure health status. It was developed to measure health-related quality of life, estimate disease burden and compare disease-specific benchmarks across populations. The VR-12 items measure eight health domains: general health perceptions, physical functioning and role limitations due to physical and emotional problems, bodily pain, energy-fatigue, social functioning and mental health. The instrument produces a physical health and mental health. Assesses how much physical health has changed over a period of time. The VR instruments use a nine-point ordinal response choices for four items in the VR-12. These answers then contribute to the scales for role limitations due to physical and emotional problems and the physical and mental summary scores.
Time Frame: 6 weeks.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Carbon Fiber Implant | Titanium Implant
Number analyzed (Participants) | 3 | 4
units on a scale | 31.63 (3.72) | 25.53 (8.42)

9. Secondary Outcome: Veterans Rand Health Survey (VR-12)
Description: The Veterans Rand 12 Item Health Survey is a multipurpose, self-administered generic measure health status. It was developed to measure health-related quality of life, estimate disease burden and compare disease-specific benchmarks across populations. The VR-12 items measure 8 health domains: general health perceptions, physical functioning and role limitations due to physical and emotional problems, bodily pain, energy-fatigue, social functioning and mental health. Assesses how much physical health has changed over a period of time. The VR instruments use a nine-point ordinal response choices for four items in the VR-12. These answers then contribute to the scales for role limitations due to physical and emotional problems and the physical and mental summary scores. The score is based on the US average, which is 50. The score is a T-score which has a mean and standard deviation (mean of 50 has standard deviation of 10). The higher the score the healthier the individual.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Carbon Fiber Implant | Titanium Implant
Number analyzed (Participants) | 3 | 4
T-score | 48.03 (15.46) | 44.90 (1.95)

10. Secondary Outcome: Veterans Rand Health Survey (VR-12)
Description: The Veterans Rand 12 Item Health Survey is a multipurpose, self-administered generic measure health status. It was developed to measure health-related quality of life, estimate disease burden and compare disease-specific benchmarks across populations. The VR-12 items measure eight health domains: general health perceptions, physical functioning and role limitations due to physical and emotional problems, bodily pain, energy-fatigue, social functioning and mental health. Assesses how much physical health has changed over a period of time. The VR instruments use a nine-point ordinal response choices for four items in the VR-12. These answers then contribute to the scales for role limitations due to physical and emotional problems and the physical and mental summary scores. The score is based on the US average, which is 50. The score is a T-score which has a mean and standard deviation (mean of 50 has standard deviation of 10). The higher the score the healthier the individual.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Carbon Fiber Implant | Titanium Implant
Number analyzed (Participants) | 3 | 4
units on a scale | 36.03 (15.24) | 38.20 (20.92)

11. Secondary Outcome: Veterans Rand Health Survey (VR-12)
Description: as for outcome 10
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Carbon Fiber Implant | Titanium Implant
Number analyzed (Participants) | 3 | 4
units on a scale | 41.63 (16.87) | 47.83 (19.12)

12. Secondary Outcome: Veterans Rand Health Survey (VR-12)
Description: as for outcome 10
Time Frame: 18 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Carbon Fiber Implant | Titanium Implant
Number analyzed (Participants) | 3 | 4
units on a scale | 39.93 (10.75) | 40.63 (24.31)

13. Secondary Outcome: Veterans Rand Health Survey (VR-12)
Description: as for outcome 10
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Carbon Fiber Implant | Titanium Implant
Number analyzed (Participants) | 3 | 4
units on a scale | 41.08 (6.61) | 43.07 (5.12)

14. Secondary Outcome: Veterans Rand Health Survey (VR-12)
Description: as for outcome 10
Time Frame: 3 months.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Carbon Fiber Implant | Titanium Implant
Number analyzed (Participants) | 3 | 4
units on a scale | 40.20 (18.67) | 36.10 (42.47)

15. Secondary Outcome: Veterans Rand Health Survey (VR-12)
Description: as for outcome 10
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Carbon Fiber Implant | Titanium Implant
Number analyzed (Participants) | 3 | 4
units on a scale | 39.57 (8.75) | 38.40 (10.15)

16. Secondary Outcome: Veterans Rand Health Survey (VR-12)
Description: as for outcome 10
Time Frame: 12 months.
Population: The participants were not analyzed at the 18 month time point.
Arm/Group | Carbon Fiber Implant | Titanium Implant
Number analyzed (Participants) | 0 | 0

17. Secondary Outcome: Brief Pain Inventory (BPI)
Description: The BPI is a widely used, 15-item measure of pain intensity and interference with daily life. The questionnaire assesses three key pain domains: pain intensity, pain interference, and efficacy of pain treatments or medications. The BPI rapidly assesses the functional severity of pain and its impact on function. The scale range is 0 to 10. A lower score means pain does not interfere with normal activities of daily living.
Time Frame: 6 months.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Carbon Fiber Implant | Titanium Implant
Number analyzed (Participants) | 3 | 4
units on a scale | 1.38 (1.49) | 2.75 (3.54)

18. Secondary Outcome: Veterans Rand Health Survey (VR-12) (Optional)
Description: as for outcome 8
Time Frame: 18 months.
Population: The Carbon Fiber implants (3 participants) and the Titanium implants (4 participants) were healed and did not participate in this evaluation.
Arm/Group | Carbon Fiber Implant | Titanium Implant
Number analyzed (Participants) | 0 | 0

19. Secondary Outcome: Brief Pain Inventory (BPI)
Description: The BPI is a widely used, 15-item measure of pain intensity and interference with daily life. The questionnaire assesses three key pain domains: pain intensity, pain interference, and efficacy of pain treatments or medications. The BPI rapidly assesses the functional severity of pain and its impact on function.The BPI rapidly assesses the functional severity of pain and its impact on function. The scale range is 0 to 10. A lower score means pain does not interfere with normal activities of daily living.
Time Frame: 6 months.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Carbon Fiber Implant | Titanium Implant
Number analyzed (Participants) | 3 | 4
units on a scale | 1.38 (1.49) | 2.75 (3.54)

20. Secondary Outcome: Brief Pain Inventory (BPI)
Description: The BPI is a widely used, 15-item measure of pain intensity and interference with daily life. The questionnaire assesses three key pain domains: pain intensity, pain interference, and efficacy of pain treatments or medications. The BPI rapidly assesses the functional severity of pain and its impact on function. The BPI rapidly assesses the interference of pain and its impact on function. The scale range is 0 to 10. A lower score means pain does not interfere with normal activities of daily living.
Time Frame: 6 months.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Carbon Fiber Implant | Titanium Implant
Number analyzed (Participants) | 3 | 4
units on a scale | 2.21 (0.69) | 3.10 (5.36)

21. Secondary Outcome: Brief Pain Inventory (BPI)
Description: as for outcome 20
Time Frame: 12 months.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Carbon Fiber Implant | Titanium Implant
Number analyzed (Participants) | 3 | 4
units on a scale | 3.10 (2.40) | 2.33 (4.04)

22. Secondary Outcome: Brief Pain Inventory (BPI)
Description: The BPI is a widely used, 15-item measure of pain intensity and interference with daily life. The questionnaire assesses three key pain domains: pain intensity, pain interference, and efficacy of pain treatments or medications. The BPI rapidly assesses the functional severity of pain and its impact on function. The BPI rapidly assesses the functional severity of pain and its impact on function. The scale range is 0 to 10. A lower score means pain does not interfere with normal activities of daily living.
Time Frame: 12 months.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Carbon Fiber Implant | Titanium Implant
Number analyzed (Participants) | 3 | 4
units on a scale | 1.17 (1.26) | 0.58 (0.80)

23. Secondary Outcome: Treatment Cost
Description: Compare 2 year treatment cost per patient, associated with fixation of tibial shaft fractures using novel carbon fiber implants in comparison with titanium implants. A Carbon Fiber Implant had a cost of $2,848.35 per device, as the number value below in the Outcome Measure Data Table. We were unable to obtain the cost of the Titanium Nail.
Time Frame: Baseline to 18 months.
Population: Costs were determined for 1 carbon fiber implant. Costs were not available for 2 carbon fiber implant participants and 4 Titanium implant participants.
Measure: Number; unit: Dollars
Arm/Group | Carbon Fiber Implant | Titanium Implant
Number analyzed (Participants) | 1 | 0
Dollars | 2,848.35 |

ADVERSE EVENTS:
Time Frame: Baseline through 12 months
Arm/Group | Carbon Fiber Implant | Titanium Implant
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/4
Serious Adverse Events (participants affected / at risk) | 1/3 | 0/4
Other Adverse Events (participants affected / at risk) | 0/3 | 0/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Carbon Fiber Implant (N=3) | Titanium Implant (N=4)
Right tibia malunion (Surgical and medical procedures) | 1 (1) | 0 (0)
Fracture-left proximal tibial plateau (Surgical and medical procedures) | 1 (1) | 0 (0)
Sepsis secondary to hardware infection (Infections and infestations) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-26): https://cdn.clinicaltrials.gov/large-docs/41/NCT03382041/Prot_SAP_000.pdf